CLINICAL TRIAL: NCT02573350
Title: A Phase 2, Multi-center, Uncontrolled, Open-label Trial to Evaluate Safety, Tolerability, and Efficacy of Orally Administered OPC-67683 as 100 mg BID With Optional Titration to 200 mg BID for up to Six Months Exposure in Patients With Pulmonary Multi-drug Resistant Tuberculosis
Brief Title: A Trial to Evaluate Safety, Tolerability, and Efficacy of Orally Administered OPC-67683
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 242-07-208; 2008-005107-26 (EudraCT Number)
Record Dates: First submitted 2015-09-29; First posted 2015-10-09 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-09

CONDITIONS: Tuberculosis, Multidrug-Resistant
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — OPC-67683

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Delamanid 100 mg BID + OBR (Experimental): Participants received Delamanid 100 milligrams (mg) (2x50 mg tablets), orally, twice daily (BID) along with at least 4 additional anti-TB medications per optimized background regimen (OBR) from Week 0 to Week 26. Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment.
  Interventions: Drug: Delamanid; Drug: OBR
- Delamanid 200 mg BID + OBR (Experimental): Participants received Delamanid 200 mg (4x50 mg tablets), orally, BID along with at least 4 additional anti-TB medications per OBR up to Week 26. Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment. A participant might have been titrated to Delamanid 200 mg BID after an initial hospitalization of 2 weeks. Participants were grouped according to the longest duration of Delamanid dose administered during the study.
  Interventions: Drug: Delamanid; Drug: OBR

INTERVENTIONS:
Drug: Delamanid — Delamanid was administered orally twice daily as 50-mg tablets under fed conditions in the morning and evening.
  Other Names: OPC-67683; Deltyba
Drug: OBR — Selection and administration of the treatment medications (i.e. OBRs) was based on World Health Organization (WHO's) Guidelines for the programmatic management of drug-resistant TB, in conjunction with national TB program guidelines. Study investigators could change OBR for a participant based on his/her tolerability and drug susceptibility testing (DST) results.

SUMMARY:
A phase 2, multicenter, uncontrolled, open-label trial in participants with Multi-drug Resistant Tuberculosis (MDR-TB). Only participants who completed Trial 242-07-204 (NCT00685360) were eligible. The trial was performed globally at 14 sites qualified to treat MDR-TB. All 434 participants who completed Trial 242-07-204 were eligible for this trial if there was still potential clinical benefit to them and all inclusion criteria and no exclusion criteria were met.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all trial-related procedures
* Male or female participants aged between 18 and 64 years, inclusive, at the time of enrollment into the 242-07-204 trial. Participants who were 64 years at the time of 204 enrollment and who are now 65 years, are eligible for this trial.
* Participants who have completed trial 242-07-204
* Participants judged by the investigator to have the potential for clinical benefit from OPC-67683 exposure
* Able to produce sputum for mycobacterial culture or able to obtain sputum produced through induction
* Female participants of childbearing potential must have a negative urine pregnancy test and agree to use a highly effective method of birth control throughout the participation in the trial and for 22 weeks after last dose.
* Male participants must agree to use an adequate method of contraception (double barrier) throughout the participation in the trial and for 30 weeks after last dose.

Exclusion Criteria:

* Greater than 30 days has elapsed from the participant's date of completion in the 242-07-204 trial or greater than 30 days has elapsed since the patient's trial investigator's site was initiated in this trial, whichever is later.
* A history of allergy to any nitro-imidazoles or nitro-imidazole derivates at any time.
* Use of the medications in Section 5.4.7 including: use of amiodarone at any time during the previous 12 months, use of other anti-arrhythmics for the previous 30 days, and use of certain other medications, including certain anti-depressants, anti-histamines, and macrolides, for the previous 14 days.
* Any current serious concomitant conditions or renal impairment characterized by serum creatinine levels ≥265 moles per liter (mol/L) or hepatic impairment characterized by Alanine aminotransferase (ALT) and/or aspartate transferase (AST) levels 3 times the upper limit of the laboratory reference range from the screening lab results.
* Current clinically relevant changes in the electrocardiogram (ECG) (between Trial 242-07-204 Day 56 assessment and baseline) such as any atrioventricular (AV) block, prolongation of the QRS complex over 120 milliseconds (msec) (in both male and female participants), or the corrected QT interval using Fridericia's method (QTcF) interval over 450 msec in male participants and 470 msec in female participants.
* Current clinically relevant cardiovascular disorders such as heart failure, coronary artery disease, uncontrolled or poorly controlled hypertension, arrhythmia, tachyarrhythmia or status after myocardial infarction.
* Any participants with known or reported significant psychiatric history.
* For participants with human immunodeficiency virus (HIV) infection, CD4 cell count less than 350/cubic millimeter (mm^3) or on treatment with antiretroviral medication for HIV infection.
* Karnofsky score under 50 percent (%) while hospitalized and less than 60% while not hospitalized.
* Any current diseases or conditions in which the use of nitro-imidazoles or nitro-imidazole derivates is contra-indicated.
* Evidence of clinically significant metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
* Known or suspected alcohol abuse, that is, abuse sufficient enough to compromise the safety or cooperation of the participants in the opinion of the investigator.
* Administered an investigational medicinal product (IMP) within 1 month prior to Visit 1 other than OPC-67683 given as IMP in trial 242-07-204.
* Pregnant, breast-feeding, or planning to conceive or father a child within the timeframe described in the informed consent form.
* Recent use of methadone, benzodiazepines, cocaine, amphetamine/methamphetamine, tetrahydrocannabinol, barbiturates, and opiates as determined by a urine drug screen, unless evidence is provided that the positive drug screen is the result of authorized medications or products prescribed by a physician for a non-abuse related indication.
* Any disorder that in the judgment of the investigator makes the participant not a good candidate for the trial or may prevent the participant from reliably participating in the entire course of the trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2009-03-26 (Actual); Primary Completion 2011-10-27 (Actual); Study Completion 2011-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Beijing Chest Hospital, Beijing, China
- Estonia (2):
  - North Estonian Medical Centre Foundation Center of Pulmonology, Tallinn
  - Tartu University Lung Hospital, Tartu
- State Agency of Tuberculosis and Lung Disease, Riga, Latvia
- Hospital Nacional Sergio E. Bernales, Lima, Peru
- Tropical Disease Foundation, Makati City, Philippines
- South Korea (2):
  - Younsei University Medical Center, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in the Philippines, Latvia, Estonia, South Korea, Peru, China, and Japan from 26 March 2009 to 27 October 2011.
Pre-assignment Details: The study consisted of a Pre-treatment, Treatment, and Follow-up Period. The Pre-treatment Period consisted of a screening and baseline visit. This was followed by a 26-week Treatment Period. There was also a Follow-up Period (28 to 32 days) for the collection of Adverse events (AEs).
Groups:
- Delamanid 100 mg BID + OBR: Participants received Delamanid 100 milligrams (mg) (2x50 mg tablets), orally, twice daily (BID) along with at least 4 additional anti-TB medications per optimized background regimen (OBR) from Week 0 to Week 26. Participants were administered OBR as directed by the given investigator based on World Health Organization (WHO) guidelines and clinical judgment.
Period: Overall Study
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Started | 137 | 76
Efficacy Analysis Population (Efficacy Analysis Population included all enrolled participants who had a baseline and a post-baseline measurement available for assessment of any efficacy endpoint.) | 132 | 73
Safety Population (Safety Population included all participants treated with at least one dose of Delamanid in this study.) | 137 | 76
Completed | 121 | 67
Not Completed | 16 | 9
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 3 | 4
Not completed — Subject met Withdrawal Criteria | 1 | 1
Not completed — Subject was Withdrawn from Participation by the Investigator | 3 | 1
Not completed — Subject withdrew consent to participate | 6 | 1
Not completed — Protocol Deviation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Groups:
- Delamanid 100 mg BID + OBR: Participants received Delamanid 100 mg (2x50 mg tablets), orally, BID along with at least 4 additional anti-TB medications per OBR from Week 0 to Week 26. Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment.
- Total: Total of all reporting groups
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Total
Number analyzed (Participants) | 137 | 76 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (12.36) | 37.1 (10.98) | 36.9 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 21 | 62
  Male | 96 | 55 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 17 | 39
  Not Hispanic or Latino | 115 | 59 | 174
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 100 | 24 | 124
  Race: White | 16 | 34 | 50
  Race: Other | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Abnormality in Vital Signs
Description: Vital signs included weight (kg), body temperature (degree Celsius), heart rate [beats/minute (bpm)], systolic and diastolic blood pressure [millimetre of mercury (mm Hg)]. The criteria for clinically significant abnormal value for: weight was decrease or increase of >=5% in body weight, heart rate was <=60 bpm and decrease of >=15 bpm; >=120 bpm and Increase of >=15 bpm, systolic blood pressure (SBP) <=90 mm Hg and decrease of >=20 mm Hg; diastolic blood pressure (DBP) <=50 mm Hg and decrease of >=15 mm Hg, all vital signs relative to Baseline. Baseline is Study 204 completion visit (Day 84) for participants who complete the baseline visit within 7 days of completing Study 204. Only categories with data for potentially clinically significant abnormal vital sign parameter values are reported.
Time Frame: From first dose of study drug up to Week 26
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants
  Weight Decrease of >=5%: number analyzed (Participants) | 133 | 72
  Weight Decrease of >=5% | 23 | 11
  Weight Increase of >=5%: number analyzed (Participants) | 133 | 72
  Weight Increase of >=5% | 34 | 25
  Heart Rate: <=60 bpm and Decrease of >=15 bpm: number analyzed (Participants) | 133 | 72
  Heart Rate: <=60 bpm and Decrease of >=15 bpm | 10 | 11
  Heart Rate: >=120 bpm and Increase of >=15 bpm: number analyzed (Participants) | 133 | 72
  Heart Rate: >=120 bpm and Increase of >=15 bpm | 1 | 0
  SBP: <=90 mm Hg and Decrease of >=20 mm Hg: number analyzed (Participants) | 133 | 72
  SBP: <=90 mm Hg and Decrease of >=20 mm Hg | 16 | 2
  SBP: >=160 mm Hg and Increase of >=20 mm Hg: number analyzed (Participants) | 133 | 72
  SBP: >=160 mm Hg and Increase of >=20 mm Hg | 3 | 0
  DBP: <=50 mm Hg and Decrease of >=15 mm Hg: number analyzed (Participants) | 133 | 72
  DBP: <=50 mm Hg and Decrease of >=15 mm Hg | 1 | 2

2. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Values
Description: The criteria for clinically significant abnormal ECG values were ventricular rate outlier (<50 bpm and decrease of >=25%, >100 bpm and increase of >=25%), PR outlier (increase of >=25% when PR >200 milliseconds (ms)), QRS outlier (increase of >=25% when QRS >100 ms), QT (new onset (in treatment period but not at Baseline) [>500 ms]), QT interval corrected by Bazett's formula (QTcB) (new onset [>450, >480, >500 ms], increase of >=30 ms and <= 60 ms or increase of >60 ms), QT interval corrected by Fridericia's formula (QTcF) (new onset [>450, >480, >500 ms], increase of >=30 ms and <= 60 ms or increase of >60 ms), new abnormal U waves, new ST segment changes, new T wave changes, new abnormal rhythm, new conduction abnormality were reported as categories. Only categories with data are reported.
Time Frame: From first dose of study drug up to Week 26
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants
  QRS Outlier | 2 | 0
  QT Interval, New Onset (>500 msec) | 1 | 0
  QTcB Interval, New Onset (>450 msec) | 62 | 37
  QTcB Interval, New Onset (>480 msec) | 11 | 7
  QTcB Interval, New Onset (>500 msec) | 2 | 3
  QTcB Interval, Increase from Baseline >=30 msec and <=60 msec | 58 | 39
  QTcB Interval, Increase from Baseline >60 msec | 5 | 7
  QTcF Interval, New Onset (>450 msec) | 23 | 10
  QTcF Interval, New Onset (>480 msec) | 3 | 1
  QTcF Interval, New Onset (>500 msec) | 1 | 1
  QTcF Interval, Increase from Baseline >=30 msec and <=60 msec | 36 | 30
  QTcF Interval, Increase from Baseline >60 msec | 4 | 4
  Ventricular Rate Notable Changes, <50 bpm and Decrease from Baseline of >=25% | 1 | 2
  Ventricular Rate Notable Changes, >100 bpm and Increase from Baseline of >=25% | 16 | 8
  New Abnormal U Waves | 4 | 0
  New ST Segment Changes | 11 | 2
  New T Waves Changes | 27 | 14
  New Abnormal Rhythm | 44 | 22
  New Conduction | 10 | 4

3. Primary Outcome: Number of Participants With Clinical Significant Abnormality in Laboratory Test
Description: Laboratory assessments included parameters for serum chemistry (alkaline phosphatase, alanine aminotransferase, alanine transaminase, total bilirubin, cholesterol, gamma-glutamyl transferase, glucose, lactic dehydrogenase, potassium, sodium, triglycerides, uric acid), hematology (white blood cell count eosinophils, absolute, hematocrit, hemoglobin, lymphocytes, absolute, mean corpuscular volume, neutrophil, bands, neutrophils, neutrophils, absolute, platelet count, red blood cell (RBC) count, reticulocyte count) and urinalysis (blood, epithelial cast, granular cast, hyaline cast, RBCs per high power field (RBC/HPF)). The participants were categorized based on the clinically significant laboratory values as per predefined criteria. The categories with at least one participant with clinically significant value outside the normal range for laboratory assessments are reported.
Time Frame: From first dose of study drug up to Week 26
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study. Number analyzed is the number of participants with at least one post-baseline result for the given test.
Measure: Count of Participants; unit: Participants
Groups:
- Delamanid 200 mg BID + OBR: Participants received delamanid 200 mg (4x50 mg tablets), orally, BID plus OBR up to Week 26. Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment. A participant may have been titrated to delamanid 200 mg BID after an initial hospitalization of 2 weeks. Participants were grouped according to the longest duration of delamanid dose administered during the study.
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants
  Alkaline Phosphatase: number analyzed (Participants) | 136 | 76
  Alkaline Phosphatase | 0 | 1
  Alanine Aminotransferase (SGPT) | 2 | 1
  Aspartate Aminotransferase (SGOT) | 2 | 1
  Total Bilirubin | 7 | 4
  Cholesterol | 1 | 2
  GAMMA-Glutamyl Transferase | 2 | 2
  Glucose: number analyzed (Participants) | 136 | 76
  Glucose | 5 | 3
  Lactic Dehydrogenase | 22 | 5
  Potassium | 13 | 10
  Sodium | 16 | 16
  Triglycerides | 9 | 3
  Uric Acid: number analyzed (Participants) | 136 | 76
  Uric Acid | 9 | 8
  Eosinophils, Absolute: number analyzed (Participants) | 130 | 76
  Eosinophils, Absolute | 10 | 3
  Hematocrit | 2 | 4
  Hemoglobin | 61 | 24
  Lymphocytes, Absolute | 0 | 1
  Mean Corpuscular Volume | 20 | 13
  Neutrophil, Bands: number analyzed (Participants) | 28 | 30
  Neutrophil, Bands | 0 | 1
  Neutrophils | 6 | 2
  Neutrophils, Absolute | 17 | 10
  Platelet Count | 5 | 3
  Red Blood Cell Count | 15 | 14
  Reticulocyte Count | 9 | 5
  White Blood Count | 6 | 3
  Blood Urine Present | 41 | 29
  Epithelial Cast in Urine: number analyzed (Participants) | 1 | 1
  Epithelial Cast in Urine | 1 | 1
  Granular Cast in Urine: number analyzed (Participants) | 9 | 3
  Granular Cast in Urine | 9 | 3
  Hyaline Cast in Urine: number analyzed (Participants) | 6 | 7
  Hyaline Cast in Urine | 6 | 6
  RBC/HPF in Urine: number analyzed (Participants) | 13 | 5
  RBC/HPF in Urine | 13 | 5

4. Primary Outcome: Number of Participants With Abnormality in Audiometry at Baseline
Description: Audiometry assessments were done at Baseline.
Time Frame: Baseline
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants | 90 | 34

5. Primary Outcome: Number of Participants With Abnormality in Visual Acuity
Time Frame: From first dose of study drug up to Week 26
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants | 45 | 35

6. Primary Outcome: Number of Participants With Abnormality in Neurological and Psychiatric Assessment Reported as Treatment-emergent Adverse Event (TEAE)
Description: Participants with abnormal neurological and psychiatric assessments were reported. An adverse event (AE) is any untoward medical occurrence in a participant/clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with treatment. A TEAE is any new AE or worsening of an existing condition after initiation of study drug.
Time Frame: From first dose through 28 days after last dose of study drug (up to approximately 30 weeks)
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants
  Neurological Disorders | 63 | 25
  Psychiatric Disorders | 44 | 38

7. Primary Outcome: Number of Participants With Clinical Significant Abnormality in Thyroid Function Test Reported as TEAE
Description: Participants with abnormal thyroid free T4 nanograms per deciliter (ng/dL) and thyroid-stimulating hormone (>=3 OR <=0.3 micro-international units per litre (uIU/mL). An AE is any untoward medical occurrence in a participant/clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with treatment. A TEAE is any new AE or worsening of an existing condition after initiation of study drug.
Time Frame: From first dose through 28 days after last dose of study drug (up to approximately 30 weeks)
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Delamanid 100mg BID + OBR: Participants received Delamanid 100 mg (2x50 mg tablets), orally, BID along with at least 4 additional anti-TB medications per OBR from Week 0 to Week 26. Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment.
- Delamanid 200mg BID + OBR: Participants received Delamanid 200 mg (4x50 mg tablets), orally, BID along with at least 4 additional anti-TB medications per OBR up to Week 26. Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment. A participant might have been titrated to Delamanid 200 mg BID after an initial hospitalization of 2 weeks. Participants were grouped according to the longest duration of Delamanid dose administered during the study.
Arm/Group | Delamanid 100mg BID + OBR | Delamanid 200mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants | 0 | 1

8. Primary Outcome: Number of Participants With Any Concomitant Medication Usage
Description: Concomitant medications are defined as medications that started on or after the first day of study treatment or were started prior to study treatment but were ongoing on the first day of study treatment.
Time Frame: From first dose of study drug up to Week 26
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants | 135 | 75

9. Primary Outcome: Percentage of Participants With At Least One TEAEs and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant/clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with treatment. A TEAE is any new AE or worsening of an existing condition after initiation of study drug. An SAE is an AE that resulted in death, inpatient hospitalization/prolongation of existing hospitalization, persistent or significant disability or incapacity, life-threatening, a congenital anomaly/birth defect, or an important medical event.
Time Frame: From first dose through 28 days after last dose of study drug (up to approximately 30 weeks)
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 137 | 76
percentage of participants
  TEAEs | 92.0 | 97.4
  SAEs | 13.9 | 7.9

10. Primary Outcome: Number of Participants With Clinical Significant Abnormality in Coagulation (PT and aPTT) Reported as TEAE
Description: Participants with clinically significant abnormal coagulation (prothrombin time (PT) >17.5 seconds and activated partial thromboplastin time (aPTT) >45 seconds) were reported.
Time Frame: From first dose through 28 days after last dose of study drug (up to approximately 30 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid 100mg BID + OBR | Delamanid 200mg BID + OBR
Number analyzed (Participants) | 137 | 76
Participants
  Activated Partial Thromboplastin Time | 12 | 8
  Prothrombin Time: number analyzed (Participants) | 122 | 42
  Prothrombin Time | 2 | 1

11. Primary Outcome: Number of Participants With Clinical Significant Abnormality in Cortisol
Description: Participants with clinically significant cortisol >=26 micrograms/decilitre (ug/dL) were reported.
Time Frame: From first dose of study drug up to Week 26
Population: Safety Population included all participants treated with at least one dose of Delamanid in this study. Overall number of participants analyzed is the number of participants with at least one post-baseline result for the given test.
Measure: Count of Participants; unit: Participants
Arm/Group | Delamanid 100mg BID + OBR | Delamanid 200mg BID + OBR
Number analyzed (Participants) | 136 | 76
Participants | 44 | 19

12. Secondary Outcome: Percentage of Treatment Responders Using the Mycobacterial Growth Indicator Tube (MGIT) Culture System
Description: Treatment Responder was defined as a participant classified as sustained converter or a new converter. Sustained Converter was defined as a participant with sputum culture conversion (SCC) at baseline and without any positive culture result during the 26-week trial period. New converter was defined as a participant without SCC at baseline who subsequently met the definition of SCC. A participant was classified as having achieved SCC if he/she achieved 2 consecutive sputum cultures negative for growth of mycobacterium tuberculosis (MTB) at least 28 days apart after his/her last sputum culture that was positive for growth. The total percentage of treatment responders was calculated as the number of sustained converters plus the number of new converters divided by the total number of participants in the analysis population. Efficacy was assessed by the MGIT sputum culture system (ie, sputum culture conversion).
Time Frame: Week 26
Population: Efficacy Analysis Population included all enrolled participants who had a baseline and a post-baseline measurement available for assessment of any efficacy endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 79.5 [71.7 to 86.1] | 75.3 [63.9 to 84.7]

13. Secondary Outcome: Percentage of Treatment Responders Using Solid Culture Medium
Description: Treatment Responder was defined as a participant classified as sustained converter or a new converter. Sustained Converter was defined as a participant with SCC at baseline and without any positive culture result during the 26-week trial period. New converter was defined as a participant without SCC at baseline who subsequently met the definition of SCC. A participant was classified as having achieved SCC if he/she achieved 2 consecutive sputum cultures negative for growth of MTB at least 28 days apart after his/her last sputum culture that was positive for growth. The total percentage of treatment responders was calculated as the number of sustained converters plus the number of new converters divided by the total number of participants in the analysis population. Efficacy was assessed by the solid culture medium (ie, sputum culture conversion)
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 81.8 [74.2 to 88.0] | 82.2 [71.5 to 90.2]

14. Secondary Outcome: Percentage of Treatment Non-responders Using the MGIT Culture System
Description: Non-responders were defined as participants classified as non-converter or reverter. Non-converters were defined as participants without SCC at baseline and who did not achieve SCC during the 26-week trial period whereas reverters were participants with SCC at baseline and at least one positive post-baseline result. The total percentage of treatment non-responders was calculated as the number of reverters plus the number of non-converters divided by the total number of participants in the analysis population. Efficacy was assessed by the MGIT sputum culture system (ie, sputum culture conversion)
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 20.5 [13.9 to 28.3] | 24.7 [15.3 to 36.1]

15. Secondary Outcome: Percentage of Treatment Non-responders Using Solid Culture Medium
Description: Non-responders were defined as participants classified as non-converter or reverter. Non-converters were defined as participants without SCC at baseline and who did not achieve SCC during the 26-week trial period whereas reverters were participants with SCC at baseline and at least one positive post-baseline result. Treatment Non-responders was calculated as the number of reverters plus the number of non-converters divided by the total number of participants in the analysis population. Efficacy was assessed by the Solid culture medium (ie, sputum culture conversion).
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 18.2 [12.0 to 25.8] | 17.8 [9.8 to 28.5]

16. Secondary Outcome: Percentage of Sustained Converters Using the MGIT Culture System
Description: The total percentage of sustained converters was defined as the percentage of participants in the analysis dataset who had SCC at baseline and non-positive sputum culture results for all post-baseline visits. Efficacy was assessed by the MGIT sputum culture system (ie, sputum culture conversion)
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 69.7 [61.1 to 77.4] | 69.9 [58.0 to 80.1]

17. Secondary Outcome: Percentage of Sustained Converters Using Solid Culture Medium
Description: The total percentage of sustained converters was defined as percentage of participants in the analysis dataset who had SCC at baseline and non-positive sputum culture results for all post-baseline visits. Determined by Solid culture medium. Efficacy was assessed by the solid culture medium (ie, sputum culture conversion)
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 74.2 [65.9 to 81.5] | 72.6 [60.9 to 82.4]

18. Secondary Outcome: Percentage of New Converters Using the MGIT Culture System
Description: The total percentage of new converters was defined as the percentage of participants in the analysis dataset without SCC at baseline who achieved SCC during the 26-week trial period. Efficacy was assessed by the MGIT sputum culture system (ie, sputum culture conversion).
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 9.8 [5.3 to 16.3] | 5.5 [1.5 to 13.4]

19. Secondary Outcome: Percentage of New Converters Using Solid Culture Medium
Description: The total percentage of new converters was defined as the percentage of participants in the analysis dataset without SCC at baseline who achieved SCC during the 26-week trial period. Efficacy was assessed by the solid culture medium (ie, sputum culture conversion).
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 7.6 [3.7 to 13.5] | 9.6 [3.9 to 18.8]

20. Secondary Outcome: Percentage of Non-converters Using the MGIT Culture System
Description: The total percentage of non-converters was defined as the percentage of participants in the analysis dataset without SCC at baseline and who did not achieve SCC during the 26-week trial period. Efficacy was assessed by the MGIT sputum culture system (ie, sputum culture conversion).
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 8.3 [4.2 to 14.4] | 13.7 [6.8 to 23.8]

21. Secondary Outcome: Percentage of Non-converters Using Solid Culture Medium
Description: The total percentage of non-converters was defined as the percentage of participants in the analysis dataset without SCC at baseline and who did not achieve SCC during the 26-week trial period. Efficacy was assessed by the solid culture medium (ie, sputum culture conversion).
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 6.8 [3.2 to 12.5] | 9.6 [3.9 to 18.8]

22. Secondary Outcome: Percentage of Reverters Using the MGIT Culture System
Description: The total percentage of reverters was defined as the percentage of participants in the analysis dataset with SCC at baseline and at least one positive post-baseline result. Efficacy was assessed by the MGIT sputum culture system (ie, sputum culture conversion).
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 12.1 [7.1 to 18.9] | 11.0 [4.9 to 20.5]

23. Secondary Outcome: Percentage of Reverters Using Solid Culture Medium
Description: The total percentage of reverters was defined as the percentage of participants in the analysis dataset with SCC at baseline and at least one positive post-baseline result. Efficacy was assessed by the solid culture medium (ie, sputum culture conversion).
Time Frame: Week 26
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 11.4 [6.5 to 18.0] | 8.2 [3.1 to 17.0]

24. Secondary Outcome: Percentage of Participants Who Developed Resistance to Delamanid While on Treatment
Description: Resistance was defined as mycobacterium tuberculosis (MTB) growth on the delamanid-containing medium of greater than 1% of that on the drug-free medium. The overall resistance to delamanid during the study was assessed.
Time Frame: Up to Week 26
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 132 | 73
percentage of participants | 1.5 | 2.7

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose of study drug (up to approximately 30 weeks)
Description: Safety Population included all participants treated with at least one dose of Delamanid in this study.
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
All-Cause Mortality (participants affected / at risk) | 1/137 | 0/76
Serious Adverse Events (participants affected / at risk) | 19/137 | 6/76
Other Adverse Events (participants affected / at risk) | 126/137 | 73/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delamanid 100 mg BID + OBR (N=137) | Delamanid 200 mg BID + OBR (N=76)
Right ventricular failure (Cardiac disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Appendicitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pulmonary tuberculoma (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 2 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Electrocardiogram Qt prolonged (Investigations) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Delamanid 100 mg BID + OBR (N=137) | Delamanid 200 mg BID + OBR (N=76)
Palpitations (Cardiac disorders) | 18 | 0
Tinnitus (Ear and labyrinth disorders) | 16 | 5
Abdominal pain (Gastrointestinal disorders) | 8 | 1
Abdominal pain lower (Gastrointestinal disorders) | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 19 | 6
Diarrhoea (Gastrointestinal disorders) | 14 | 7
Dyspepsia (Gastrointestinal disorders) | 7 | 6
Gastritis (Gastrointestinal disorders) | 10 | 8
Nausea (Gastrointestinal disorders) | 20 | 15
Toothache (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 24 | 5
Chest pain (General disorders) | 12 | 6
Hyperbilirubinaemia (Hepatobiliary disorders) | 8 | 1
Folliculitis (Infections and infestations) | 1 | 4
Lung infection (Infections and infestations) | 7 | 2
Nasopharyngitis (Infections and infestations) | 12 | 12
Pharyngitis (Infections and infestations) | 6 | 4
Tracheobronchitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 11 | 5
Blood cortisol increased (Investigations) | 12 | 1
Decreased appetite (Metabolism and nutrition disorders) | 11 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 2
Dizziness (Nervous system disorders) | 19 | 3
Headache (Nervous system disorders) | 42 | 12
Paraesthesia (Nervous system disorders) | 8 | 5
Somnolence (Nervous system disorders) | 14 | 4
Tremor (Nervous system disorders) | 9 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 7
Anxiety (Psychiatric disorders) | 6 | 7
Depression (Psychiatric disorders) | 4 | 4
Insomnia (Psychiatric disorders) | 30 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 11 | 2
Hot flush (Vascular disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.